CLINICAL TRIAL: NCT01137149
Title: Behavioral Activation Therapy With Adolescents
Brief Title: Behavioral Activation With Depressed Adolescents
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Elizabeth McCauley, PHD, Seattle Childrens' Hospital/University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BA Adolescent Study
Record Dates: First submitted 2010-06-01; First posted 2010-06-04 (Estimated); Last update posted 2010-06-04 (Estimated); Status verified 2010-06

CONDITIONS: Depression
Keywords: Adolescent Depression; Treatment of depression in adolescents; Behavioral activation treatment for depressed adolescents
MeSH Terms: conditions — Depression | interventions — Behavior Therapy; Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment as Usual- Psychotherapy (Active Comparator): The TAU condition will be implemented consistent with usual and customary clinical practices within the Child Psychiatry Clinic at Seattle Children's Hospital (SCH. Within the SCH system, TAU for a depressed adolescent will typically consist of an individual therapy approach with adjunct family sessions and pharmacotherapy as deemed necessary by the primary therapist. The therapeutic approach typically used is cognitive behavioral but is administered in an eclectic, non-manualized fashion. Therapists for the TAU arm of the study will be care providers currently working within the SCH system. For this phase of the study, we will draw on clinicians whose level of experience is comparable to that of the Behavioral Activation therapists.
  Interventions: Behavioral: Treatment as Usual- Psychotherapy
- Behavioral Acitivation Therapy (Experimental): Behavioral activation is a 12 week psychotherapeutic intervention utilizing a semi-structured format. Initial sessions focus on specific areas (Assessment and orientation, Activation, Problem Solving, Goal Setting, Overcoming Barriers, Avoidance) interspersed as needed by sessions that focus on individual issues and applications. In these sessions the therapists maintains the session structure, but can use techniques presented in earlier sessions based on their functional analysis of the particular case. Parents participate in at least two of the ATA sessions but more active parental participation can be included as needed.
  Interventions: Behavioral: Behavioral Activation Therapy

INTERVENTIONS:
Behavioral: Behavioral Activation Therapy — Behavioral activation is a 12 week psychotherapeutic intervention utilizing a semi-structured format. Initial sessions focus on specific areas (Assessment and orientation, Activation, Problem Solving, Goal Setting, Overcoming Barriers, Avoidance) interspersed as needed by sessions that focus on individual issues and applications. In these sessions the therapists maintains the session structure, but can use techniques presented in earlier sessions based on their functional analysis of the particular case. Parents participate in at least two of the ATA sessions but more active parental participation can be included as needed.
  Other Names: Behavioral Therapy
  Arms: Behavioral Acitivation Therapy
Behavioral: Treatment as Usual- Psychotherapy — The TAU condition will be implemented consistent with usual and customary clinical practices within the Child Psychiatry Clinic at Seattle Children's Hospital (SCH. Within the SCH system, TAU for a depressed adolescent will typically consist of an individual therapy approach with adjunct family sessions and pharmacotherapy as deemed necessary by the primary therapist. The therapeutic approach typically used is cognitive behavioral but is administered in an eclectic, non-manualized fashion. Therapists for the TAU arm of the study will be care providers currently working within the SCH system. For this phase of the study, we will draw on clinicians whose level of experience is comparable to that of the Behavioral Activation therapists.
  Arms: Treatment as Usual- Psychotherapy

SUMMARY:
Twenty percent of adolescents will have at least one episode of clinical depression by age 18, and 65% will experience transient or less severe depressive symptoms. Depression compromises the process of adolescent development by interfering with academic, occupational, and social functioning, and increasing risk for substance use and suicide. Although initial research provides some support for both pharmacological and psychosocial interventions, many depressed teens do not respond to these interventions, and others experience a relapse of symptoms within one year. Furthermore, concerns about antidepressant medications increasing suicide risk have raised additional caution about use of pharmacotherapy with adolescents. As such, the importance of developing innovative treatment options for depressed adolescents is critical. Cognitive Behavioral Therapy (CBT) has been demonstrated to be effective in the treatment of depressed adults, with more modest efficacy data when used with children and adolescents. Interestingly, recent data from the adult literature suggests the positive outcomes of CBT can be achieved and surpassed by interventions that are purely behavioral in nature. Behavioral interventions may be easier to implement with many adolescents and may provide a better developmental fit for depressed adolescents. The present project proposes to develop a manualized Behavioral Activation (BA) Therapy for depressed adolescents, test its adaptability, acceptability, and feasibility in an open clinical trial with 12 adolescents (aged 12-17), and following further treatment refinement, test its efficacy in a randomized controlled trial of 50 adolescents (aged 12-17), in which 25 will be randomized to BA Therapy and 25 will receive "Treatment as Usual (TAU)." In this randomized controlled trial, depressed adolescents will receive 12-weeks of BA Therapy or TAU. Psychiatric and psychosocial functioning will be assessed at the beginning, middle, and end of treatment. A naturalistic follow-up will be conducted 4 and 9 months post-treatment. Assuming that BA will outperform "usual" approaches to therapy with depressed youth, the data will provide the basis for the development of a larger randomized controlled trial comparing the efficacy of BA against other widely studied approaches to the treatment of depression in youth, namely pharmacotherapy in the form of Selective Serotonin Reuptake Inhibitors (SSRIs), and CBT.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 11 and 18;
2. one parent/legal guardian willing to participate in the study;
3. primary diagnosis of a depressive disorder (Major Depressive Disorder, Dysthymia, Depression NOS);
4. Short Mood and Feelings Questionnaire >11;
5. Children's Depression Rating Scale score > 45;
6. willingness to be randomized into either treatment group.

Exclusion Criteria:

Adolescents will be excluded if they meet any of the following criteria:

1. primary diagnosis other than a depressive disorder;
2. presence of psychotic and/or manic symptoms;
3. presence of chronic medical condition;
4. presence of active substance abuse/dependence;
5. presence of chronic self-mutilation or cutting (e.g., persistent, severe, and/or requiring medical treatment);
6. presence acute or chronic suicidality (e.g., > 3 suicidal gestures in the past year),
7. previous unfavorable response to an adequate regimen of either CBT or antidepressant treatment in the prior year, and/or (8)developmental delay.

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2006-10; Primary Completion 2011-01 (Estimated); Study Completion 2011-01 (Estimated)

PRIMARY OUTCOMES:
Children's Depression Rating Scale-Revised (CDRS-R) | Baseline assessment
  The CDRS-R, an interview-based measure, will be administered by the blind independent evaluator with both the parent and adolescent. The CDRS-R has been found to be a sensitive and reliable severity measure of depression in children and adolescents. Ratings are made across 17 symptoms, including depressed feelings, sleep disturbance, and suicidal ideation, on a scale of 1 (no difficulties) to 7 (severe clinically significant difficulties). A raw score at or above 45 or a T-score at or above 65 is reported to be increasingly indicative of a likely depressive disorder.
Children's Depression Rating Scale-Revised (CDRS-R) | End of Active Treatment (12 weeks)
  The CDRS-R, an interview-based measure, will be administered by the blind independent evaluator with both the parent and adolescent. The CDRS-R has been found to be a sensitive and reliable severity measure of depression in children and adolescents. Ratings are made across 17 symptoms, including depressed feelings, sleep disturbance, and suicidal ideation, on a scale of 1 (no difficulties) to 7 (severe clinically significant difficulties). A raw score at or above 45 or a T-score at or above 65 is reported to be increasingly indicative of a likely depressive disorder.
Children's Depression Rating Scale-Revised (CDRS-R) | At 9 months Follow-up Evaluaton
  The CDRS-R, an interview-based measure, will be administered by the blind independent evaluator with both the parent and adolescent. The CDRS-R has been found to be a sensitive and reliable severity measure of depression in children and adolescents. Ratings are made across 17 symptoms, including depressed feelings, sleep disturbance, and suicidal ideation, on a scale of 1 (no difficulties) to 7 (severe clinically significant difficulties). A raw score at or above 45 or a T-score at or above 65 is reported to be increasingly indicative of a likely depressive disorder.

SECONDARY OUTCOMES:
Clinical Global Impressions Scale | Baseline (severity) assessment
  The Clinical Global Impressions Scale will be utilized as an assessment of the severity of the adolescent's symptoms/level of symptom improvement as rated by the independent clinical evaluator. Scores range on a scale from 1-7, with lower scores denoting better outcome. The CGI measure has been widely utilized in a number of treatment outcome studies with adolescents to ascertain treatment response rate, with scores of 1 (very much improved) or 2 (much improved) indicating positive response to treatment.
Clinical Global Impressions Scale | At the end of active treatment (12 weeks)
  The Clinical Global Impressions Scale will be utilized as an assessment of the severity of the adolescent's symptoms/level of symptom improvement as rated by the independent clinical evaluator. Scores range on a scale from 1-7, with lower scores denoting better outcome. The CGI measure has been widely utilized in a number of treatment outcome studies with adolescents to ascertain treatment response rate, with scores of 1 (very much improved) or 2 (much improved) indicating positive response to treatment.
Clinical Global Impressions Scale | At the 9 month follow-up evaluation
  The Clinical Global Impressions Scale will be utilized as an assessment of the severity of the adolescent's symptoms/level of symptom improvement as rated by the independent clinical evaluator. Scores range on a scale from 1-7, with lower scores denoting better outcome. The CGI measure has been widely utilized in a number of treatment outcome studies with adolescents to ascertain treatment response rate, with scores of 1 (very much improved) or 2 (much improved) indicating positive response to treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth McCauley, PHD, Principal Investigator — Seattle Children's Hospital
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States